CLINICAL TRIAL: NCT03456024
Title: Chronic Abdominal Pain and Discomfort in Morbid Obese Patients Before and After Sleeve Gastrectomy
Brief Title: Abdominal Pain and Symptoms Post Gastric Sleeve
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Voss Sykehus (Unknown)
Responsible Party: Principal Investigator, Tom Mala, Consultant surgeon, phd, Oslo University Hospital
Other Study IDs: Sleeve and abdominal pain
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Abdominal Pain; Quality of Life
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questinnaire

SUMMARY:
Exploration of abdominal pain post sleeve gastrectomy in morbid obese patients

DETAILED DESCRIPTION:
The primary aim is to evaluate abdominal pain in morbid obese patients before and after sleeve gastrectomy. The investigators will especially focus on chronic abdominal pain, and its relation to quality of life and weight loss. In a sub-analysis the investigators will compare the findings of the present cohort with patients operated with Roux-en-Y gastric bypass.

Primary endpoints/outcomes:

- Define the prevalence of chronic abdominal pain 2 years after sleeve gastrectomy

Secondary endpoints/outcomes:

- Evaluate and characterise chronic abdominal pain in regard to:

* Weight development
* Obesity-related comorbidities
* Health-related quality of life
* Postoperative complications
* Metabolic effects after surgery
* Nutritional status
* Socioeconomic status

ELIGIBILITY:
* Inclusion criteria

  * Patients undergoing sleeve gastrectomy at the Center for Morbid Obesity and Bariatric Surgery, Oslo University Hospital and a collaborating center.
  * Signed written and informed consent for study enrollment
* Exclusion criteria

  * Patients who dont understand Norwegian language
  * Previous bariatric surgery
  * Indication for sleeve gastrectomy for other reasons than for morbid obesity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients scheduled for sleeve gastrectomy for morbid obesity at Oslo University Hospital and Voss sykehus
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-11-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic abdominal pain 2 years after gastric sleeve | 2 years
  questionnaire

SECONDARY OUTCOMES:
Quality of life related to abdominal pain and symptoms | 2 years
  questionnaire (SF-36v2, OP scale)

OTHER OUTCOMES:
Comparison to gastric bypass | 2 year
  questionnaire (SF36v2, OP scale)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Mala, MD,Phd, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided